CLINICAL TRIAL: NCT01234350
Title: A Prospective Observational Safety Study in Patients With Advanced Prostate Cancer Treated With FIRMAGON (Degarelix) or a GnRH Agonist
Brief Title: A Safety Study in Patients With Advanced Prostate Cancer Treated With FIRMAGON
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE200486 CS39
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- FIRMAGON
- GnRH Agonist

SUMMARY:
This study is a large observational study, set-up to observe how long-term treatment with FIRMAGON (hormone regulator) compare to other treatments in regards to cardiovascular events, changes in bone density, changes in blood sugar levels or liver enzyme levels in subjects with prostate cancer. Subjects will be treated according to their routine clinical care and not dictated by the study. As the study is observational in nature, the study will collect data relating to the events specified above. Subjects that agree to this study will be followed-up for 5 years. Subject data will be collected every 3 months for the first 2 years and every 6 months for the last 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer and indicated for androgen deprivation therapy (ADT)
* Decision made to prescribe ADT prior to enrolment
* Willing and able to provide written informed consent

Exclusion Criteria:

* Participation in an interventional clinical study in which any treatment or follow-up is mandated
* Treatment with a GnRH receptor antagonist other than FIRMAGON
* Had previous or is currently under hormonal management of prostate cancer, except for subjects who have undergone therapy with curative intention where neoadjuvant/adjuvant therapy allowed for maximum 6 months. Treatment should be terminated at least 6 months prior to baseline.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with prostate cancer from primary care
Sampling Method: Non-Probability Sample
Enrollment: 1493 (Actual)
Dates: Start 2011-01; Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (160):
- Belgium (17):
  - Onze-Lieve-Vrouwziekenhuis, Aalst
  - Ziekenhuisnetwerk Antwerpen - AZ Stuivenberg, Antwerp
  - AZ Sint-Jan AV, Bruges
  - Hôpitaux IRIS Sud, Brussels
  - Université Catholique de Louvain, Brussels
  - Hôpital Erasme, Bruxelle
  - AZ Sint-Blasius, Dendermonde
  - AZ Jan Palfijn, Ghent
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - UZ Gent, Ghent
  - Regionaal Ziekenhuis Jan Yperman VZW, Ieper
  - AZ Groeninge - Campus Sint-Maarten, Kortrijk
  - CHU de Liège, Liège
  - Centre Hospitalier Universitaire Ambroise Paré, Mons
  - AZ Damiaan, Ostend
  - AZ-Sint-Elizabeth VZW, Zottegem
- Denmark (6):
  - Aalborg Sygehus, Aalborg
  - Rigshospitalet, Copenhagen
  - Fredericia Hospital, Sygehus Lillebaelt, Fredericia
  - Herlev Hospital, Herlev
  - Holstebro Sygehus, Holstebro
  - Regionhospitalet Viborg, Viborg
- Finland (6):
  - Docrates clinic, Helsinki
  - Pohjois-Karjalan keskussairaala, Joensuu
  - Seinäjoen keskussairaala, Seinäjoki
  - Tampereen yliopistollinen sairaala, Tampere
  - Turun yliopistollinen keskussairaala, Turku
  - Peijaksen sairaala, Vantaa
- France (27):
  - CHRU Angers, Angers
  - Centre Hospitalier d'Athis Mons site Caron, Athis-Mons
  - Hopital Tenon, Aubervilliers
  - Clinique Rhone Durance, Avignon
  - CHU Saint-Jacques, Besançon
  - Centre Hospitalier Laennec, Clermont-Ferrand
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Ramsay Sante, Évry
  - Groupement hospitalier Edouard Herriot, Lyon
  - Cabinet Médical 65 prado, Marseille
  - CHU Nord, Marseille
  - Hopital de la Conception, Marseille
  - Polyclinique Saint-Jean, Melun
  - Clinique du Pont de Chaume, Montauban
  - Clinique Beausoleil, Montpellier
  - Centre d'Urologie de Nancy, Nancy
  - Hôpital Max Fourestier, Nanterre
  - Centre Hospitalier Georges Renon, Niort
  - Groupe hospitalo-universitaire Caremeau, Nîmes
  - Hopital Tenon, Paris
  - Clinique du Ter, Ploemeur
  - Clinic De L'Europe, Pontoise
  - Hopital Pontchaillou, Rennes
  - Clinique Saint Michel, Toulon
  - Clinique St Jean Languedoc, Toulouse
  - Hopital Bretonneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy
- Germany (22):
  - Gemeinschaftspraxis Dres Effert und Benedic, Aachen
  - Praxis Dr. Schlichter, Bad Bergzaben
  - Praxis Dr. Markus Hentschel, Bautzen
  - Praxis Dr. Richter, Bonn
  - Urologie im Schlosscarree, Braunschweig
  - Praxis Dr. Ahmad Haider, Bremerhaven
  - Praxis Dr. Krieger, Chemnitz
  - Urologie Chemnitz, Chemnitz
  - Praxis Dr. Thomas Harms, Cologne
  - Gemeinschaftspraxis fur Urologie, Dachau
  - Klinikpraxis fur Urologie, Dinslaken
  - Praxis Dr. Schönfelder, Hamburg
  - Gemeinschaftspraxis Urologie, Kiel
  - Urologische Gemeinschaftspraxis, Kiel
  - Gemeinshaftspraxis Rudolph & Wörner, Kirchheim
  - Vituro, Leipzig
  - Praxis Alexander von Keitz, Marburg
  - Praxis Dr. Peczat, Nienburg
  - Studienzentrum München-Planegg, Planegg
  - Urologische Gemeinschaftspraxis, Reutlingen
  - Praxis Dr. Jan Franz, Tostedt
  - Praxis fur Urologie, Wuppertal
- Greece (21):
  - "Agios Savas" Anticancer-Oncology Hospital of Athens, Athens
  - "G. Gennimtas" General Hospital of Athens, Athens
  - "Laiko" General Hospital of Athens, Athens
  - Amalia Fleming General Hospital of Athens, Athens
  - Errikos Dynan Hospital of Athens, Athens
  - Eurokliniki Hospital of Athens, Athens
  - Evaggelismos General Hospital, Athens
  - General Hospital of Athens "Ag. Olga" - Konstantopouleion, Athens
  - Ippokrateio Hospital of Athens, Athens
  - Korgialenio-Benakio, Athens
  - Pe. Pa.G.N:I Hospital, Heraklion
  - General hospital of Kalamata, Kalamata
  - IASO General Hospital, Kalamata
  - University Hospital of Larissa, Larissa
  - Aghios Andreas General Hospital of Patras, Pátrai
  - University General Hospital of Patras, Pátrai
  - General Hospital of Piraeus "Tzanneio", Piraeus
  - "G. Gennimtas" General Hospital of Thessaloniki, Thessaloniki
  - 2nd IKA-ETAM "Panagia" General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Volos "Achillopouleio", Volos
- Hungary (6):
  - Azarka Zsuzsanna és Társa Bt, Budapest
  - UROFOR Bt, Debrecen
  - Kiskunhalasi Semmelweis Kórház Kht., Kiskunhalas
  - Miskolci Semmelweis Ignác Egészségügyi Központ és Egyetemi Oktató Kórház Nonprofit Kft, Miskolc
  - Uro-Clin Kft, Pécs
  - FEjér Megyei Szent György Kórhaz, Székesfehérvár
- Ireland (3):
  - Beacon Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University College Hospital, Galway
- Italy (13):
  - Medical Consulting Center S.r.l., Avellino
  - Azienda Sanitaria Regionale del Molise (ASREM), Campobasso
  - Azienda Ospedaliera Mater Domini di Catanzaro, Catanzaro
  - Azienda Ospedaliera Carlo Poma, Mantova
  - Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliera Monaldi, Napoli
  - Azienda Sanitaria Locale Salerno, Nocera Inferiore
  - Ospedale Santa Maria delle Croci, Ravenna
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - Azienda Ospedaliera Universitaria OO.RR. S.Giovanni di Dio e Ruggi d'Aragona, Salerno
  - ASL 4 di Teramo, Teramo
  - Ospedale "San Pio da Pietrelcina", Vasto
- Netherlands (5):
  - AMC, Amsterdam
  - Catharina ziekenhuis, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Diaconessenhuis Leiden, Leiden
  - MC Haaglanden, The Hague
- Norway (5):
  - Vestre Viken HF, Sykehuset Asker og Baerum, Asker
  - Haukeland Universitetssykehus, Bergen
  - Helse Nordmore og Romsdal HF, Kristiansund Sykehus, Kristiansund
  - Olso Universitetssykehus HF, Radiumhospitalet, Oslo
  - Oslo Universitetssykehus, Aker, Oslo
- Portugal (3):
  - Clinica de Santo Antonio, Lisbon
  - Hospital Militar, Lisbon
  - Hospital Santa Maria, Lisbon
- Slovakia (18):
  - VEBMED, s.r.o., Bošany
  - CUIMED, s.r.o., Bratislava
  - Nemocnica Svateho Michala, a.s., Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - URO clinic, s.r.o., Bratislava
  - Poliklinika Galanta, Galanta
  - MEDICONA s.r.o., Košice
  - UROCENTRUM LEVICE, s.r.o., Levice
  - Poliklinika Malacky, Malacky
  - Univerzitna nemocnica Martin, Martin
  - UROEXAM, spol. s r.o., Nitra
  - CENTRUM UROLOGIE Povazska Bystrica s.r.o, Považská Bystrica
  - MILAB, s.r.o., Prešov
  - Nemocnica s poliklinikou Skalica, a.s., Skalica
  - UROCENTRUM SALA, s.r.o., Šaľa
  - M & M & M, s.r.o., Topoľčany
  - PRIVATNA UROLOGICKA AMBULANCIA s.r.o., Trenčín
  - UROREX, s.r.o., Vráble
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Urozentrum Zürich, Zurich
- United Kingdom (6):
  - Homerton University Hospital, London
  - Kings College Hospital, London
  - Royal Marsden Hospital, London
  - Whipps Cross Hospital, London
  - East Surrey Hospital, Redhill
  - Sunderland Royal Hospital, Sunderland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 136 sites in 15 European countries (Belgium, Denmark, Finland, France, Germany, Greece, Hungary, Ireland, Italy, Netherlands, Norway, Portugal, Slovakia, Switzerland, United Kingdom) recruited subjects to this observational study between January 2011 to April 2013, and the last subject completed the last visit in March 2018.
Pre-assignment Details: A total of 1,515 subjects were screened, of which 1,493 subjects were found to be eligible and exposed to treatment; 1,000 subjects in the FIRMAGON group and 493 subjects in the gonadotrophin releasing hormone (GnRH) agonist group.
Groups:
- FIRMAGON: FIRMAGON (Degarelix, a GnRH antagonist) was prescribed in accordance with the approved label
- GnRH Agonist: Any GnRH agonist prescribed in accordance with the approved labels
Period: Overall Study
Arm/Group | FIRMAGON | GnRH Agonist
Started | 1000 | 493
Completed | 313 | 226
Not Completed | 687 | 267
Not completed — Adverse Event | 277 | 92
Not completed — Withdrawal by Subject | 61 | 36
Not completed — Lost to Follow-up | 115 | 47
Not completed — Covers a diverse set of reasons | 234 | 92

BASELINE CHARACTERISTICS:
Population: The safety analysis set comprised of all subjects treated with at least one dose of medicinal product. The data was restricted to main treatment period (from signing of informed consent and administration of first dose until loss to follow-up, change/discontinuation in androgen deprivation therapy [ADT], or end-of-study visit, whatever came first).
Groups:
- Total: Total of all reporting groups
Arm/Group | FIRMAGON | GnRH Agonist | Total
Number analyzed (Participants) | 1000 | 493 | 1493
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed differs from the overall population as age was not recorded for some of the subjects.
  years
    Age: number analyzed (Participants) | 999 | 493 | 1492
    Age | 71.9 (8.33) | 73.2 (8.27) | 72.4 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1000 | 493 | 1493
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was not recorded for some subjects.
  Participants
    number analyzed (Participants) | 780 | 385 | 1165
    Hispanic or Latino | 12 | 5 | 17
    Not Hispanic or Latino | 697 | 353 | 1050
    Unknown or Not Reported | 71 | 27 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed differs from the overall population as race was not recorded for some of the subjects.
  Participants
    number analyzed (Participants) | 780 | 385 | 1165
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 14 | 23
    White | 745 | 360 | 1105
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 26 | 8 | 34
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number analyzed differs from the overall population as baseline body mass index (BMI) was not calculated for some of the subjects.
  kg/m^2
    number analyzed (Participants) | 786 | 406 | 1192
    (all) | 27 (3.91) | 26.8 (3.82) | 26.9 (3.88)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Adverse Events of Special Interest (AESI): Cardiovascular Events
Description: The incidence rate (IR) expressed as number of events per 100 patient-years of exposure (PYE).
Time Frame: From baseline upto 5 years (every 3 months from the first 2 years of the study; every 6 months for the last 3 years of the study)
Population: The safety analysis set comprised of all subjects treated with at least one dose of medicinal product. The data was restricted to main treatment period (from signing of informed consent and administration of first dose until loss to follow-up, change/discontinuation in ADT, or end-of-study visit, whatever came first).
Measure: Number; unit: Events per 100 PYE
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
Events per 100 PYE | 3.8 | 4.5
Statistical Analysis 1: Comparison: FIRMAGON vs GnRH Agonist; The IRs were estimated using a Poisson-mixture regression model; Test type: Other; p = 0.4007, Wald test — Poisson-mixture regression was used to model the influence of age, stage of disease, and relevant medical history along with the treatment group effect on the number of events adjusted for individual study exposures measured in 100 PYE; The IRs for each treatment arm with 95% confidence interval (CI), and incidence rate ratio (IRRs) with 95% CI and p-values were based on Wald test; IRR = 0.829, 95% CI 2-sided [0.536 to 1.283] — IRR for treatment with the lower 95% confidence limit >1 suggest increased risk of AESI; upper confidence limit <1 suggest decreased risk of AESI with the use of FIRMAGON. The limit including 1 suggests no difference b/w treatment groups

2. Primary Outcome: Incidence Rate of AESI: Decreased Bone Density
Description: IR of osteoporosis or osteopenia and bone fracture events are presented. The IR is expressed as number of events per 100 PYE.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Events per 100 PYE
Groups:
- GnRH Agonist: Any GnRH prescribed in accordance with the approved labels
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
Events per 100 PYE
  Osteoporosis or Osteopenia | 1.1 | 1.4
  Bone fracture | 0.3 | 0.1
Statistical Analysis 1: Comparison: FIRMAGON vs GnRH Agonist; For osteoporosis and osteopenia events. The IRs were estimated using Poisson-mixture regression model; Test type: Other; p = 0.6710, Wald test — [p-value comment as in outcome 1, analysis 1]; The IRs for each treatment arm with 95% CI, and IRRs with 95% CI and p-values were based on Wald test; IRR = 0.874, 95% CI 2-sided [0.470 to 1.626] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FIRMAGON vs GnRH Agonist; For bone fracture events. The IRs were estimated using Poisson-mixture regression model; Test type: Other; p = 0.4544, Wald test — [p-value comment as in outcome 1, analysis 1]; The IRs for each treatment arm with 95% CI, and IRRs with 95% CI and p-values were based on Wald test; IRR = 1.857, 95% CI 2-sided [0.367 to 9.403] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Incidence Rate of AESI: Glucose Intolerance or Type 2 Diabetes Mellitus (T2DM)
Description: IR of new onset or exacerbation of glucose intolerance or T2DM were presented. The IR expressed as number of events per 100 PYE.
  Glucose intolerance events were defined as events of levels of fasting glucose of 6.1 to 6.9 mmol/L
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Events per 100 PYE
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
Events per 100 PYE
  Glucose intolerance | 15.3 | 13.2
  T2DM | 1.8 | 0.7
Statistical Analysis 1: Comparison: FIRMAGON vs GnRH Agonist; For glucose intolerance. The IRs were estimated using Poisson-mixture regression model; Test type: Other; p = 0.2529, Wald test — Poisson mixture regression was used to model the influence of age, stage of disease, and history of diabetes mellitus along with the treatment group effect on the number of events adjusted for individual study exposures measured in 100 PYE; The IRs for each treatment arm with 95% CI, and IRRs with 95% CI and p-values were based on Wald test; IRR = 1.193, 95% CI 2-sided [0.882 to 1.613] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FIRMAGON vs GnRH Agonist; For T2DM. The IRs were estimated using Poisson-mixture regression model; Test type: Other; p = 0.0208, Wald test — Poisson-mixture regression is used to model the influence of age, stage of disease, and relevant medical history along with the treatment group effect on the number of events adjusted for individual trial exposures measured in 100 PYE; The IRs for each treatment arm with 95% CI, and IRRs with 95% CI and p-values were based on Wald test; IRR = 2.623, 95% CI 2-sided [1.158 to 5.944] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Change in Hepatic Enzymes
Description: Change from baseline in hepatic enzyme levels (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and alkaline phosphatase [ALP]) are presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: IU/L
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
IU/L
  ALT (Visit 2, Month 3): number analyzed (Participants) | 302 | 120
  ALT (Visit 2, Month 3) | 0.1 [-70 to 63] | 0.1 [-19 to 82]
  ALT (Visit 3, Month 6): number analyzed (Participants) | 272 | 115
  ALT (Visit 3, Month 6) | 0.1 [-65 to 174] | 0.1 [-41 to 125]
  ALT (Visit 4, Month 9): number analyzed (Participants) | 243 | 109
  ALT (Visit 4, Month 9) | 0.0 [-66 to 55] | 0.0 [-22 to 54]
  ALT (Visit 5, Month 12): number analyzed (Participants) | 212 | 109
  ALT (Visit 5, Month 12) | 0.0 [-63 to 57] | 0.0 [-38 to 49]
  ALT (Visit 6, Month 15): number analyzed (Participants) | 195 | 107
  ALT (Visit 6, Month 15) | -0.1 [-69 to 30] | 0.0 [-44 to 37]
  ALT (Visit 7, Month 18): number analyzed (Participants) | 183 | 98
  ALT (Visit 7, Month 18) | -0.1 [-68 to 41] | 0.1 [-26 to 77]
  ALT (Visit 8, Month 21): number analyzed (Participants) | 170 | 99
  ALT (Visit 8, Month 21) | -0.1 [-70 to 204] | 0.1 [-25 to 49]
  ALT (Visit 9, Month 24): number analyzed (Participants) | 155 | 97
  ALT (Visit 9, Month 24) | -0.1 [-65 to 332] | 0.0 [-24 to 20]
  ALT (Visit 10, Month 30): number analyzed (Participants) | 151 | 89
  ALT (Visit 10, Month 30) | -0.1 [-80 to 28] | 0.0 [-23 to 26]
  ALT (Visit 11, Month 36): number analyzed (Participants) | 134 | 89
  ALT (Visit 11, Month 36) | -0.1 [-50 to 317] | 0.0 [-16 to 90]
  ALT (Visit 12, Month 42): number analyzed (Participants) | 123 | 73
  ALT (Visit 12, Month 42) | -0.1 [-35 to 31] | 0.0 [-44 to 33]
  ALT (Visit 13, Month 48): number analyzed (Participants) | 95 | 66
  ALT (Visit 13, Month 48) | -1.0 [-36 to 97] | 0.0 [-45 to 28]
  ALT (Visit 14, Month 54): number analyzed (Participants) | 79 | 56
  ALT (Visit 14, Month 54) | -1.0 [-53 to 32] | -0.1 [-32 to 13]
  ALT (Visit 15, end of trial [EOT], Month 60): number analyzed (Participants) | 58 | 42
  ALT (Visit 15, end of trial [EOT], Month 60) | -0.2 [-30 to 33] | 0.0 [-16 to 16]
  ALP (Visit 2, Month 3): number analyzed (Participants) | 278 | 131
  ALP (Visit 2, Month 3) | 0.0 [-661 to 738] | -0.1 [-632 to 240]
  ALP (Visit 3, Month 6): number analyzed (Participants) | 247 | 123
  ALP (Visit 3, Month 6) | 0.0 [-990 to 979] | 0.0 [-649 to 135]
  ALP (Visit 4, Month 9): number analyzed (Participants) | 223 | 116
  ALP (Visit 4, Month 9) | 0.0 [-1009 to 1024] | 0.1 [-658 to 225]
  ALP (Visit 5, Month 12): number analyzed (Participants) | 203 | 111
  ALP (Visit 5, Month 12) | 0.0 [-1029 to 614] | 0.1 [-661 to 184]
  ALP (Visit 6, Month 15): number analyzed (Participants) | 181 | 113
  ALP (Visit 6, Month 15) | 0.1 [-1027 to 957] | 0.0 [-225 to 370]
  ALP (Visit 7, Month 18): number analyzed (Participants) | 184 | 105
  ALP (Visit 7, Month 18) | 0.1 [-1031 to 475] | 0.1 [-217 to 889]
  ALP (Visit 8, Month 21): number analyzed (Participants) | 156 | 109
  ALP (Visit 8, Month 21) | 0.0 [-539 to 777] | 0.0 [-197 to 364]
  ALP (Visit 9, Month 24): number analyzed (Participants) | 148 | 104
  ALP (Visit 9, Month 24) | 0.1 [-756 to 307] | 0.1 [-228 to 446]
  ALP (Visit 10, Month 30): number analyzed (Participants) | 139 | 96
  ALP (Visit 10, Month 30) | 0.0 [-540 to 300] | 0.1 [-211 to 169]
  ALP (Visit 11, Month 36): number analyzed (Participants) | 122 | 96
  ALP (Visit 11, Month 36) | -0.3 [-764 to 748] | 0.1 [-185 to 386]
  ALP (Visit 12, Month 42): number analyzed (Participants) | 113 | 84
  ALP (Visit 12, Month 42) | -0.1 [-773 to 1238] | 0.2 [-182 to 235]
  ALP (Visit 13, Month 48): number analyzed (Participants) | 84 | 70
  ALP (Visit 13, Month 48) | -0.1 [-785 to 657] | 0.2 [-204 to 114]
  ALP (Visit 14, Month 54): number analyzed (Participants) | 80 | 69
  ALP (Visit 14, Month 54) | -0.2 [-779 to 79] | 0.3 [-197 to 104]
  ALP (Visit 15 [EOT], Month 60): number analyzed (Participants) | 57 | 54
  ALP (Visit 15 [EOT], Month 60) | -5.0 [-756 to 164] | 0.2 [-157 to 89]
  AST (Visit 2, Month 6): number analyzed (Participants) | 290 | 126
  AST (Visit 2, Month 6) | 0.1 [-72 to 64] | 0.0 [-82 to 49]
  AST (Visit 3, Month 9): number analyzed (Participants) | 256 | 121
  AST (Visit 3, Month 9) | 0.1 [-73 to 79] | 0.0 [-74 to 37]
  AST (Visit 4, Month 12): number analyzed (Participants) | 233 | 113
  AST (Visit 4, Month 12) | 0.0 [-68 to 69] | 0.1 [-41 to 60]
  AST (Visit 5, Month 15): number analyzed (Participants) | 202 | 115
  AST (Visit 5, Month 15) | 0.0 [-72 to 44] | 0.1 [-77 to 108]
  AST (Visit 6, Month 15): number analyzed (Participants) | 188 | 108
  AST (Visit 6, Month 15) | 0.0 [-73 to 194] | 0.1 [-78 to 54]
  AST (Visit 7, Month 18): number analyzed (Participants) | 169 | 104
  AST (Visit 7, Month 18) | 0.0 [-72 to 108] | 0.1 [-37 to 60]
  AST (Visit 8, Month 21): number analyzed (Participants) | 161 | 103
  AST (Visit 8, Month 21) | 0.0 [-73 to 25] | 0.1 [-45 to 73]
  AST (Visit 9, Month 24): number analyzed (Participants) | 143 | 95
  AST (Visit 9, Month 24) | 0.0 [-75 to 68] | 0.0 [-43 to 32]
  AST (Visit 10, Month 30): number analyzed (Participants) | 136 | 92
  AST (Visit 10, Month 30) | 0.0 [-73 to 28] | 0.0 [-46 to 665]
  AST (Visit 11, Month 36): number analyzed (Participants) | 124 | 92
  AST (Visit 11, Month 36) | 0.0 [-72 to 57] | 0.1 [-43 to 43]
  AST (Visit 12, Month 40): number analyzed (Participants) | 113 | 76
  AST (Visit 12, Month 40) | 0.0 [-70 to 21] | 0.0 [-53 to 30]
  AST (Visit 13, Month 48): number analyzed (Participants) | 90 | 68
  AST (Visit 13, Month 48) | -0.1 [-70 to 167] | 0.0 [-52 to 18]
  AST (Visit 14, Month 54): number analyzed (Participants) | 73 | 54
  AST (Visit 14, Month 54) | -0.3 [-68 to 34] | 0.0 [-48 to 29]
  AST (Visit 15 [EOT], Month 60): number analyzed (Participants) | 52 | 44
  AST (Visit 15 [EOT], Month 60) | 0.0 [-35 to 22] | 0.0 [-42 to 15]

5. Primary Outcome: Change in Hepatic Enzymes
Description: Change from baseline in hepatic enzyme level (bilirubin) is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: umol/L
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
umol/L
  Visit 2, Month 3: number analyzed (Participants) | 208 | 78
  Visit 2, Month 3 | -1.0 [-169 to 97] | -1.0 [-108 to 15]
  Visit 3, Month 6: number analyzed (Participants) | 194 | 70
  Visit 3, Month 6 | -1.0 [-234 to 216] | -2.0 [-16 to 136]
  Visit 4, Month 9: number analyzed (Participants) | 168 | 65
  Visit 4, Month 9 | -0.9 [-233 to 38] | -0.6 [-18 to 93]
  Visit 5, Month 12: number analyzed (Participants) | 152 | 64
  Visit 5, Month 12 | -1.3 [-98 to 113] | -0.6 [-285 to 13]
  Visit 6, Month 15: number analyzed (Participants) | 137 | 67
  Visit 6, Month 15 | -0.9 [-22 to 166] | -0.7 [-23 to 245]
  Visit 7, Month 18: number analyzed (Participants) | 131 | 57
  Visit 7, Month 18 | -1.2 [-99 to 111] | -0.4 [-28 to 65]
  Visit 8, Month 21: number analyzed (Participants) | 125 | 61
  Visit 8, Month 21 | -1.5 [-200 to 145] | -1.1 [-287 to 12]
  Visit 9, Month 24: number analyzed (Participants) | 111 | 54
  Visit 9, Month 24 | -0.8 [-196 to 141] | -1.5 [-113 to 15]
  Visit 10, Month 30: number analyzed (Participants) | 103 | 56
  Visit 10, Month 30 | -1.4 [-199 to 14] | -0.4 [-282 to 126]
  Visit 11, Month 36: number analyzed (Participants) | 88 | 50
  Visit 11, Month 36 | -1.8 [-200 to 137] | -3.2 [-282 to 11]
  Visit 12, Month 40: number analyzed (Participants) | 81 | 47
  Visit 12, Month 40 | -1.6 [-196 to 129] | -1.7 [-112 to 10]
  Visit 13, Month 48: number analyzed (Participants) | 62 | 45
  Visit 13, Month 48 | -0.9 [-192 to 58] | -1.9 [-286 to 125]
  Visit 14, Month 54: number analyzed (Participants) | 56 | 37
  Visit 14, Month 54 | -1.3 [-98 to 145] | -1.9 [-286 to 83]
  Visit 15 (EOT), Month 60: number analyzed (Participants) | 43 | 30
  Visit 15 (EOT), Month 60 | -1.9 [-101 to 14] | -0.8 [-286 to 13]

6. Primary Outcome: Change in Serum Glucose
Description: Change from baseline in serum glucose are presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: mmol/L
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
mmol/L
  Visit 2, Month 3: number analyzed (Participants) | 225 | 89
  Visit 2, Month 3 | 0.0 [-5 to 9] | 0.0 [-5 to 6]
  Visit 3, Month 6: number analyzed (Participants) | 202 | 89
  Visit 3, Month 6 | 0.0 [-6 to 4] | 0.0 [-11 to 7]
  Visit 4, Month 9: number analyzed (Participants) | 183 | 83
  Visit 4, Month 9 | 0.1 [-7 to 14] | 0.1 [-7 to 5]
  Visit 5, Month 12: number analyzed (Participants) | 166 | 91
  Visit 5, Month 12 | 0.0 [-8 to 6] | 0.0 [-14 to 9]
  Visit 6, Month 15: number analyzed (Participants) | 158 | 79
  Visit 6, Month 15 | 0.0 [-6 to 5] | 0.2 [-8 to 6]
  Visit 7, Month 18: number analyzed (Participants) | 149 | 83
  Visit 7, Month 18 | 0.0 [-8 to 3] | 0.2 [-13 to 6]
  Visit 8, Month 21: number analyzed (Participants) | 146 | 79
  Visit 8, Month 21 | 0.0 [-9 to 5] | 0.1 [-12 to 6]
  Visit 9, Month 24: number analyzed (Participants) | 129 | 76
  Visit 9, Month 24 | 0.0 [-6 to 4] | -0.2 [-4 to 6]
  Visit 10, Month 30: number analyzed (Participants) | 123 | 74
  Visit 10, Month 30 | 0.0 [-6 to 4] | 0.0 [-8 to 7]
  Visit 11, Month 36: number analyzed (Participants) | 114 | 71
  Visit 11, Month 36 | 0.0 [-6 to 4] | 0.2 [-5 to 9]
  Visit 12, Month 42: number analyzed (Participants) | 103 | 52
  Visit 12, Month 42 | 0.1 [-6 to 4] | -0.1 [-4 to 2]
  Visit 13, Month 48: number analyzed (Participants) | 78 | 51
  Visit 13, Month 48 | 0.2 [-3 to 8] | 0.0 [-6 to 6]
  Visit 14, Month 54: number analyzed (Participants) | 66 | 48
  Visit 14, Month 54 | 0.0 [-5 to 3] | 0.1 [-10 to 9]
  Visit 15 (EOT), Month 60: number analyzed (Participants) | 52 | 37
  Visit 15 (EOT), Month 60 | 0.1 [-1 to 9] | 0.2 [-10 to 3]

7. Secondary Outcome: Number and Classification of New Adverse Drug Reactions (ADRs)
Description: An ADR was defined as an AE assessed by investigator as possibly/probably related to the investigational product. Any new potentially unrecognized ADRs were presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: New ADR
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
New ADR | 0 | 0

8. Secondary Outcome: Long Term Evaluation of Clinical Evolution of Prostate Cancer
Description: Change in prostate specific antigen (PSA) is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
ng/mL
  Visit 2, Month 3: number analyzed (Participants) | 709 | 348
  Visit 2, Month 3 | -20.1 [-788 to 297] | -10.7 [-438 to 160]
  Visit 3, Month 6: number analyzed (Participants) | 657 | 358
  Visit 3, Month 6 | -19.1 [-789 to 161] | -11.4 [-466 to 399]
  Visit 4, Month 9: number analyzed (Participants) | 625 | 326
  Visit 4, Month 9 | -17.0 [-788 to 583] | -11.5 [-477 to 260]
  Visit 5, Month 12: number analyzed (Participants) | 575 | 340
  Visit 5, Month 12 | -17.5 [-787 to 578] | -12.9 [-465 to 311]
  Visit 6, Month 15: number analyzed (Participants) | 526 | 318
  Visit 6, Month 15 | -15.8 [-783 to 493] | -11.0 [-472 to 648]
  Visit 7, Month 18: number analyzed (Participants) | 499 | 304
  Visit 7, Month 18 | -16.0 [-770 to 665] | -11.3 [-477 to 790]
  Visit 8, Month 21: number analyzed (Participants) | 450 | 279
  Visit 8, Month 21 | -14.4 [-770 to 201] | -11.0 [-485 to 567]
  Visit 9, Month 24: number analyzed (Participants) | 421 | 282
  Visit 9, Month 24 | -14.0 [-770 to 325] | -11.9 [-442 to 297]
  Visit 10, Month 30: number analyzed (Participants) | 395 | 270
  Visit 10, Month 30 | -14.6 [-770 to 692] | -11.7 [-488 to 394]
  Visit 11, Month 36: number analyzed (Participants) | 352 | 257
  Visit 11, Month 36 | -15.4 [-770 to 410] | -11.4 [-485 to 590]
  Visit 12, Month 42: number analyzed (Participants) | 309 | 229
  Visit 12, Month 42 | -16.7 [-770 to 548] | -10.5 [-486 to 498]
  Visit 13, Month 48: number analyzed (Participants) | 270 | 210
  Visit 13, Month 48 | -15.1 [-770 to 487] | -9.5 [-484 to 248]
  Visit 14, Month 54: number analyzed (Participants) | 246 | 192
  Visit 14, Month 54 | -13.0 [-770 to 204] | -8.9 [-482 to 98]
  Visit 15 (EOT), Month 69: number analyzed (Participants) | 177 | 145
  Visit 15 (EOT), Month 69 | -14.7 [-770 to 405] | -9.0 [-407 to 39]

9. Secondary Outcome: Changes in Testosterone Levels
Description: Change from baseline in testosterone levels are presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
ng/mL
  Visit 2, Month 3: number analyzed (Participants) | 195 | 110
  Visit 2, Month 3 | -3.6 [-38 to 33] | -3.0 [-10 to 30]
  Visit 3, Month 6: number analyzed (Participants) | 158 | 99
  Visit 3, Month 6 | -3.8 [-38 to 17] | -3.3 [-19 to 0]
  Visit 4, Month 9: number analyzed (Participants) | 155 | 94
  Visit 4, Month 9 | -3.6 [-38 to 53] | -3.190 [-10.16 to -0.03]
  Visit 5, Month 12: number analyzed (Participants) | 136 | 85
  Visit 5, Month 12 | -3.6 [-38 to 9] | -3.236 [-9.79 to 8.82]
  Visit 6, Month 15: number analyzed (Participants) | 110 | 76
  Visit 6, Month 15 | -3.5 [-38 to 10] | -3.146 [-10.16 to 0.10]
  Visit 7, Month 18: number analyzed (Participants) | 118 | 74
  Visit 7, Month 18 | -3.6 [-22 to 35] | -3.127 [-9.79 to 5.34]
  Visit 8, Month 21: number analyzed (Participants) | 91 | 73
  Visit 8, Month 21 | -3.3 [-38 to 22] | -3.175 [-9.80 to -0.03]
  Visit 9, Month 24: number analyzed (Participants) | 91 | 63
  Visit 9, Month 24 | -3.5 [-37 to 19] | -3.041 [-9.80 to 1.14]
  Visit 10, Month 30: number analyzed (Participants) | 82 | 68
  Visit 10, Month 30 | -3.5 [-22 to 2] | -2.847 [-9.78 to 3.57]
  Visit 11, Month 36: number analyzed (Participants) | 75 | 63
  Visit 11, Month 36 | -3.7 [-22 to 2] | -2.977 [-9.78 to 3.85]
  Visit 12, Month 42: number analyzed (Participants) | 69 | 52
  Visit 12, Month 42 | -3.7 [-22 to 2] | -2.835 [-9.65 to 0.13]
  Visit 13, Month 48: number analyzed (Participants) | 61 | 56
  Visit 13, Month 48 | -3.930 [-22.00 to 10.78] | -2.6 [-10 to 4]
  Visit 14, Month 54: number analyzed (Participants) | 51 | 49
  Visit 14, Month 54 | -3.380 [-22.23 to 7.35] | -2.463 [-9.61 to 3.60]
  Visit 15 (EOT), Month 60: number analyzed (Participants) | 44 | 46
  Visit 15 (EOT), Month 60 | -3.870 [-22.23 to 1.61] | -2.2 [-8 to 3]

10. Secondary Outcome: All-cause of Mortality
Description: A summary of IRs of all-cause mortality is presented.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Events per 100 PYE
Arm/Group | FIRMAGON | GnRH Agonist
Number analyzed (Participants) | 1000 | 493
Events per 100 PYE | 6.5 | 5.1
Statistical Analysis 1: Comparison: FIRMAGON vs GnRH Agonist; The analyses of all-cause mortality was based on logistic regressions; Test type: Other; p = 0.0821, Regression, Logistic — A logistic regression was used to model the influence of age, stage of disease and relevant medical history along with the treatment group on the time to event for all-cause mortality; Logistic regression was used to model the influence of age, stage of disease and relevant medical history along with the treatment group; Odds Ratio (OR) = 0.747, 95% CI 2-sided [0.537 to 1.038]

ADVERSE EVENTS:
Time Frame: From baseline upto 5 years (every 3 months from the first 2 years of the study; every 6 months for the last 3 years of the study)
Description: An AE was defined as any untoward medical occurrence in a subject participating in a clinical investigation who received a pharmaceutical product.
  The safety analysis set comprised of all subjects treated with at least one dose of medicinal product. The data was restricted to main treatment period (from signing of informed consent and administration of first dose until loss to follow-up, change/discontinuation in ADT, or end-of-study visit, whatever came first).
Arm/Group | FIRMAGON | GnRH Agonist
All-Cause Mortality (participants affected / at risk) | 141/1000 | 72/493
Serious Adverse Events (participants affected / at risk) | 236/1000 | 144/493
Other Adverse Events (participants affected / at risk) | 294/1000 | 110/493
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRMAGON (N=1000) | GnRH Agonist (N=493)
Anaemia (Blood and lymphatic system disorders) | 6 (9) | 10 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 8 (8) | 5 (5)
Myocardial infarction (Cardiac disorders) | 9 (9) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (5) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery disease (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Subventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 25 (26) | 12 (12)
Death (General disorders) | 12 (12) | 6 (6)
General physical health deterioration (General disorders) | 10 (10) | 5 (5)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 3 (3)
Asthenia (General disorders) | 3 (3) | 3 (3)
Chest pain (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 4 (5) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 9 (10)
Urinary tract infection (Infections and infestations) | 5 (5) | 6 (8)
Sepsis (Infections and infestations) | 6 (6) | 3 (3)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Echinococciasis (Infections and infestations) | 1 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Injection site abscess (Infections and infestations) | 1 (2) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Haematocrit dereased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 40 (41) | 10 (11)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hormone-refractory prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Spinal cord compression (Nervous system disorders) | 3 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesis (Nervous system disorders) | 2 (3) | 0 (0)
Anterograde amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciosness (Nervous system disorders) | 0 (0) | 1 (1)
Mobility decreased (Nervous system disorders) | 1 (1) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 12 (12) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 8 (8) | 1 (1)
Renal failure (Renal and urinary disorders) | 6 (6) | 2 (2)
Haematuria (Renal and urinary disorders) | 4 (5) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 1 (2)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (2)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney enlargement (Renal and urinary disorders) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectoprostatic fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyapnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye prosthesis insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Ileostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical induction of coma (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRMAGON (N=1000) | GnRH Agonist (N=493)
Injection site pain (General disorders) | 100 (226) | 2 (2)
Prostatic specific antigen increased (Investigations) | 80 (90) | 26 (29)
Hot flush (Vascular disorders) | 166 (172) | 88 (92)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2010-06-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT01234350/Prot_000.pdf
  • Statistical Analysis Plan (2014-08-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT01234350/SAP_001.pdf